CLINICAL TRIAL: NCT03629483
Title: Impact of Dexmedetomidine Combined With Ropivacaine for Postoperative Continuous Femoral Nerve Block on Postoperative Delirium and Long-term Oucomes in Elderly Patients After Single Knee Arthroplasty
Brief Title: Dexmedetomidine Combined With Ropivacaine for Postoperative Continuous Femoral Nerve Block
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial stopped by the sponsor because similar studies have been conducted.
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEX 20180516
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Elderly; Knee Arthroplasty; Nerve Block; Dexmedetomidine; Postoperative Delirium; Long-term Outcome
Keywords: Elderly; Knee Arthroplasty; Nerve Block; Dexmedetomidine; Postoperative Delirium; Long-term Outcome
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): For patients in the dexmedetomidine group, postoperative analgesia is provided in the form of continuous femoral nerve block. The formula contains a mixture of 0.2% ropivacaine 250 ml and 3.75 ug/kg dexmedetomidine. The analgesic pump is set to administer a continuous infusion at a rate of 5 ml/h for 48 hours (equivalent to dexmedetomidine infusion at a rate of 0.075 ug/kg/h).
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): For patients in the control group, postoperative analgesia is provided in the form of continuous femoral nerve block. The formula contains a mixture of 0.2% ropivacaine 250 ml and placebo (normal saline). The analgesic pump is set to administer a continuous infusion at a rate of 5 ml/h for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in this group receive continuous femoral nerve block analgesia for 48 hours after surgery. The formula is a mixture of 0.2% ropivacaine 250ml and 3.75 ug/kg dexmedetomidine. The analgesic pump is set to administer a continuous infusion at a rate of 5 ml/h (equivalent to a dexmedetomidine infusion at a rate of 0.075 ug/kg/h).
  Other Names: Continuous femoral nerve block with ropivacaine
  Arms: Dexmedetomidine group
Drug: Placebo — Patients in this group receive continuous femoral nerve block analgesia for 48 hours after surgery. The formula is a mixture of 0.2% ropivacaine 250 ml and placebo. The analgesic pump is set to administer a continuous infusion at a rate of 5 ml/h.
  Other Names: Continuous femoral nerve block with ropivacaine
  Arms: Control group

SUMMARY:
Delirium is common in the elderly after orthopedic surgery and is associated with worse outcomes. Continuous femoral nerve block is frequently used for postoperative analgesia after total knee arthoplasty. The investigators hypothesize that dexmedetomidine, when combined with ropivacaine for continuous femoral nerve block, can reduce the incidence of delirium and improve the long-term outcome in elderly patients after total knee arthroplasty.

DETAILED DESCRIPTION:
A growing number of elderly patients undergo total knee arthroplasty. Delirium is a common complication in these patients after surgery and is associated with worse outcomes, including prolonged hospital stay, poor functional recovery, decreased cognitive function, increased health care costs, and elevated mortality rate. Dexmedetomidine has been shown to prolong the duration of nerve block without neurotoxicity and improve postoperative sleep quality. The investigators hypothesize that dexmedetomidine, when combined with ropivacaine for continuous femoral nerve block, can reduce the incidence of delirium and improve the long-term outcome in elderly patients after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (≥ 65 years but < 90 years);
* Scheduled to undergo single total knee arthroplasty;
* Planned to receive continuous femoral nerve block for postoperative analgesia.

Exclusion Criteria:

* Refuse to participate in this study;
* Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
* Inability to communicate in the preoperative period because of coma, profound dementia or language barrier;
* Preoperative hemorrhagic disease or coagulopathy (platelet count, prothrombin time and/or activated partial thrombin time below the lower limit of normal);
* Preoperative obstructive sleep apnea (diagnosed as obstructive sleep apnea, or STOP-Bang score ≥3);
* Preoperative sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
* Severe hepatic dysfunction (Child-Pugh class C);
* Severe renal dysfunction (requirement of renal replacement therapy before surgery);
* ASA classification ≥ IV or unlikely to survive for more than 24 hours after surgery.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium during the first 3 days after surgery | The first 3 days after surgery
  Incidence of delirium during the first 3 days after surgery

SECONDARY OUTCOMES:
Daily prevalence of delirium during postoperative days 1-3 | The first 3 days after surgery
  Daily prevalence of delirium during postoperative days 1-3
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of non-delirium complications within 30 days after surgery | Up to 30 days after surgery
  Incidence of non-delirium complications within 30 days after surgery
All-cause 30-day mortality | At 30 days after surgery
  All-cause 30-day mortality
Quality of life at 30 days after surgery | At 30 days after surgery
  Quality of life at 30 days after surgery is assessed with the 12-items Short Form Health Survey (SF-12), a 12-item questionnaire that provides assessments of physical and mental health-related quality of life. The score ranges from 12 to 48, with higher score indicating better function.
Cognitive function at 30 days after surgery | At 30 days after surgery
  Cognitive function at 30 days after surgery is assessed with modified Telephone Interview for Cognitive Status (TICS-m), a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 50, with higher score indicating better function.
Overall survival within 3 years after surgery | Up to 3 years after surgery
  Overall survival within 3 years after surgery
Survival rates at the end of the 1st，2nd, and 3rd years after surgery | At the end of the 1st, 2nd, and 3rd years after surgery
  Survival rates at the end of the 1st，2nd, and 3rd years after surgery
Incidence of new-onset diseases within 3 years after surgery | Up to 3 years after surgery
  Incidence of new-onset diseases within 3 years after surgery
Quality of life at the end of the 1st, 2nd, and 3rd years after surgery: SF-12 | At the end of the 1st, 2nd, and 3rd years after surgery
  Quality of life at the end of the 1st, 2nd, and 3rd years after surgery is assessed with the 12-items Short Form Health Survey (SF-12), a 12-item questionnaire that provides assessments of physical and mental health-related quality of life. The score ranges from 12 to 48, with higher score indicating better function.
Cognitive function at the end of the 1st, 2nd, and 3rd years after surgery | At the end of the 1st, 2nd, and 3rd years after surgery
  Cognitive function at the end of the 1st, 2nd, and 3rd years after surgery is assessed with modified Telephone Interview for Cognitive Status (TICS-m), a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 50, with higher score indicating better function.

OTHER OUTCOMES:
Sedation level during postoperative days 1-3 | The first 3 days after surgery
  Sedation level during postoperative days 1-3 is assessed with the Richmond Agitation-Sedation Scale (RASS), of which the range is as follows: +4 (combative), +3 (very agitated), +2 (agitated), +1 (restless), 0 (alert and clam), -1 (drowsy), -2 (light sedation), -3 (moderate sedation), -4 (deep sedation), and -5 (unarousable).
Pain severity during postoperative days 1-3: NRS | The first 3 days after surgery
  Pain severity during postoperative days 1-3 is assessed with the Numeric Rating Scale (NRS), an 11-point pain scale where 0=no pain and 10=the most severe pain.
Sleep quality during postoperative days 1-3 | The first 3 days after surgery
  Sleep quality during postoperative days 1-3 is assessed with the Verran and Snyder-Halpern (VSH) Sleep Scale, an 8-item questionnaire that evaluate multiple aspects of sleep during the previous night. Each item is scored in a range from 0 (very bad) to 10 (very good), and the total VSH score is determined by the summation of these scores (range 0-80). A higher total VSH score indicates a better quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mu DL, Zhang DZ, Wang DX, Wang G, Li CJ, Meng ZT, Li YW, Liu C, Li XY. Parecoxib Supplementation to Morphine Analgesia Decreases Incidence of Delirium in Elderly Patients After Hip or Knee Replacement Surgery: A Randomized Controlled Trial. Anesth Analg. 2017 Jun;124(6):1992-2000. doi: 10.1213/ANE.0000000000002095. PMID 28525512
- [Background] Kalisvaart KJ, de Jonghe JF, Bogaards MJ, Vreeswijk R, Egberts TC, Burger BJ, Eikelenboom P, van Gool WA. Haloperidol prophylaxis for elderly hip-surgery patients at risk for delirium: a randomized placebo-controlled study. J Am Geriatr Soc. 2005 Oct;53(10):1658-66. doi: 10.1111/j.1532-5415.2005.53503.x. PMID 16181163
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Wang XL, Wang J, Mu DL, Wang DX. [Dexmedetomidine combined with ropivacaine for continuous femoral nerve block improved postoperative sleep quality in elderly patients after total knee arthroplasty]. Zhonghua Yi Xue Za Zhi. 2018 Mar 13;98(10):728-732. doi: 10.3760/cma.j.issn.0376-2491.2018.10.003. Chinese. PMID 29562395
- [Background] Choy WS, Lee SK, Kim KJ, Kam BS, Yang DS, Bae KW. Two continuous femoral nerve block strategies after TKA. Knee Surg Sports Traumatol Arthrosc. 2011 Nov;19(11):1901-8. doi: 10.1007/s00167-011-1510-4. Epub 2011 Apr 12. PMID 21484386
- [Background] Duarte VM, Fallis WM, Slonowsky D, Kwarteng K, Yeung CK. Effectiveness of femoral nerve blockade for pain control after total knee arthroplasty. J Perianesth Nurs. 2006 Oct;21(5):311-6. doi: 10.1016/j.jopan.2006.05.011. PMID 17027440
- [Background] Abdulatif M, Fawzy M, Nassar H, Hasanin A, Ollaek M, Mohamed H. The effects of perineural dexmedetomidine on the pharmacodynamic profile of femoral nerve block: a dose-finding randomised, controlled, double-blind study. Anaesthesia. 2016 Oct;71(10):1177-85. doi: 10.1111/anae.13603. PMID 27611039
- [Background] Brummett CM, Hong EK, Janda AM, Amodeo FS, Lydic R. Perineural dexmedetomidine added to ropivacaine for sciatic nerve block in rats prolongs the duration of analgesia by blocking the hyperpolarization-activated cation current. Anesthesiology. 2011 Oct;115(4):836-43. doi: 10.1097/ALN.0b013e318221fcc9. PMID 21666435
- [Background] Al-Metwalli RR, Mowafi HA, Ismail SA, Siddiqui AK, Al-Ghamdi AM, Shafi MA, El-Saleh AR. Effect of intra-articular dexmedetomidine on postoperative analgesia after arthroscopic knee surgery. Br J Anaesth. 2008 Sep;101(3):395-9. doi: 10.1093/bja/aen184. Epub 2008 Jun 20. PMID 18567675
- [Background] Brummett CM, Norat MA, Palmisano JM, Lydic R. Perineural administration of dexmedetomidine in combination with bupivacaine enhances sensory and motor blockade in sciatic nerve block without inducing neurotoxicity in rat. Anesthesiology. 2008 Sep;109(3):502-11. doi: 10.1097/ALN.0b013e318182c26b. PMID 18719449
- [Background] Behera BK, Puri GD, Ghai B. Patient-controlled epidural analgesia with fentanyl and bupivacaine provides better analgesia than intravenous morphine patient-controlled analgesia for early thoracotomy pain. J Postgrad Med. 2008 Apr-Jun;54(2):86-90. doi: 10.4103/0022-3859.40772. PMID 18480522
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Kosar CM, Tabloski PA, Travison TG, Jones RN, Schmitt EM, Puelle MR, Inloes JB, Saczynski JS, Marcantonio ER, Meagher D, Reid MC, Inouye SK. EFFECT OF PREOPERATIVE PAIN AND DEPRESSIVE SYMPTOMS ON THE DEVELOPMENT OF POSTOPERATIVE DELIRIUM. Lancet Psychiatry. 2014 Nov;1(6):431-436. doi: 10.1016/S2215-0366(14)00006-6. PMID 25642413
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Quinlan N, Rudolph JL. Postoperative delirium and functional decline after noncardiac surgery. J Am Geriatr Soc. 2011 Nov;59 Suppl 2:S301-4. doi: 10.1111/j.1532-5415.2011.03679.x. PMID 22091577
- [Background] Shi CM, Wang DX, Chen KS, Gu XE. Incidence and risk factors of delirium in critically ill patients after non-cardiac surgery. Chin Med J (Engl). 2010 Apr 20;123(8):993-9. PMID 20497703
- [Background] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702